CLINICAL TRIAL: NCT04407156
Title: Acute Kidney Injury In Corona Virus Infection Disease (COVID19) in United Kingdom
Brief Title: Epidemiology of Acute Kidney Injury in COVID19 Disease in United Kingdom
Status: Completed | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UHDB/2020/050
Record Dates: First submitted 2020-05-06; First posted 2020-05-29 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: COVID; AKI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: acute kidney injury — AKI in COVID positive cases

SUMMARY:
Severe Acute respiratory syndrome coronovirus (SARS-CoV-2) was first described in Wuhan in December 2019. It quickly spread to rest of the world and was declared pandemic by World health organisation. Initial case series focused on lung involvement in the form alveolar haemorrhages and respiratory failure. However, subsequently, there have been reports of kidney involvement resulting in severe acute kidney injury. However, the reported incidence from Chinese data has been less than 5% and detailed epidemiology of AKI in COVID-19 disease is lacking.

DETAILED DESCRIPTION:
On 31st December 2019, a cluster of pneumonia cases were detected in Hubei province of China where the cause was unclear. The cause for these cases was subsequently identified as a virus which was referred to as SARS-CoV-2, and the associated disease as COVID-19.This evolved rapidly into a global pandemic with first case reported in UK as early as on 30th January 2020. As of 30th April 2020, there have been 3.05 million laboratory confirmed cases world-wide with 161,145 cases in United Kingdom (UK) in 539,768 cases tested for COVID-19. The epidemiology of COVID-19 has differed in China, US and Italy which have different demographic characteristics, testing methods and different ways to curb the spread of infection which can be altered by many things, including behaviour, and the stringent social distancing measure.Though the pandemic started in China, as of 30th April 2020, it has reported only 58.32 cases per million people (pmp) as compared to United kingdom which has reported 2433.8 cases pmp. This has resulted in different epidemiology of COVID-19 and organ system involvement. Lung involvement in the form of alveolar haemorrhages and respiratory failure has been well document in patients with COVID-19 and has been focus of attention, however, other organs are also affected in COVID-19, but there has been limited information kidney involvement in COVID patients.

ELIGIBILITY:
Inclusion Criteria:

All patients who are admitted to the hospital with suspected COVID-19 infection between 1st March 2020 and 8th May 2020 and who meet following criteria will be included

1. Adult patients greater or equal to 18 years of age.
2. Swab results available for SARS CoV-19
3. Patients admitted to the hospital as per the national screening criteria

Exclusion Criteria:

The following patients will be excluded from the study

1. Paediatric patients as defined by age of <18 years of age
2. Swab results which are awaited
3. Patients on haemodialysis or peritoneal dialysis

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is hospitalised patients suspected to have SARS CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 724 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-06-07 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Acute kidney injury in COVID-19 | 7 days
  This is the proportion of patients with Acute kidney injury in COVID-19

SECONDARY OUTCOMES:
All-cause mortality in AKI patients | 7 days
  This is the number of deaths in COVID-19 AKI patients

CONTACTS AND LOCATIONS:
Overall Officials: Nitin V Kolhe, MD, Principal Investigator — University Hospitals of Derby and Burton
Locations (1):
- Derby Hospital NHS Foundation Trust, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The results will be shared with other researchers

REFERENCES:
- [Derived] Kolhe NV, Fluck RJ, Selby NM, Taal MW. Acute kidney injury associated with COVID-19: A retrospective cohort study. PLoS Med. 2020 Oct 30;17(10):e1003406. doi: 10.1371/journal.pmed.1003406. eCollection 2020 Oct. PMID 33125416